CLINICAL TRIAL: NCT01804257
Title: Event Marker Ingested To Trigger Event Recorder 3.0 Psychiatry Study (EMITTER 3.0 PSY)
Brief Title: Event Marker Ingested To Trigger Event Recorder 3.0 Psychiatry Study
Acronym: EMITTER3PSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proteus Digital Health, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); The Zucker Hillside Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EMITTER 3.0 PSY
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2013-03

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Adherence; Bipolar disorder; Cellular phone; Cloud computing; Computers; Computers, handheld; Digital health; Digital health feedback system; Ingestion Sensor; Medication adherence; Medication non-adherence; Medication nonadherence; Mobile phone; Mobile health; Patient adherence; Patient non-adherence; Patient nonadherence; Schizophrenia; Telehealth; Telemedicine; Telenursing; Wearable sensor
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digital Health Feedback System (DHFS) (Experimental): Ingestion Sensor, Wearable Sensor
  Interventions: Other: Digital Health Feedback System

INTERVENTIONS:
Other: Digital Health Feedback System — The digital health offering passively collects and records medication-taking behavior and other habits of daily living
  Other Names: Ingestible sensor; Wearable sensor

SUMMARY:
Feasibility study of using a digital health feedback system (DHFS) to monitor medication-taking and physiologic and behavioral parameters in patients with bipolar disorder or schizophrenia. Hypothesis: Using a digital health feedback system to characterize medication-taking behavior and activities of daily living is safe and tolerable in appropriately selected patients with bipolar disorder and schizophrenia.

DETAILED DESCRIPTION:
In this 4-week observational study conducted between May 2010 and May 2011 at 2 US academic clinical study sites, 12 adults with bipolar disorder and 16 adults with schizophrenia (all diagnosed according to DSM-IV criteria) utilized a digital health feedback system (DHFS). All subjects were on a stable regimen of oral medication. The DHFS utilized a digital tablet, consisting of an ingestion sensor that was embedded in a tablet containing nonpharmacologic excipients, which subjects coingested with their regularly prescribed medication.

The primary study objective was to compare the accuracy of DHFS in confirming digital tablet ingestion versus a method of directly observed ingestion; secondary aims included characterization of adherence and physiologic measures longitudinally in these cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 and ≤ 65 years of age
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria, by Structured Clinical Interview using DSM-IV SCID-I/P1, for either:

  i. Bipolar disorder I, II, or Not Otherwise Specified (NOS), or ii. Schizophrenia or schizoaffective disorder
* Clinical global impression scale-severity (CGI-S) of 3 or below
* Currently on a stable regimen of oral antimanic or antipsychotic medication for at least 3 months
* No anticipation to change or titrate the regimen in the next 28 days
* Willingness to adhere to study procedures
* Capacity to provide informed consent

Exclusion Criteria:

* Pregnancy, or women of child bearing potential who are not using a medically accepted means of contraception
* Serious suicide or homicide risk, as assessed by evaluating clinician
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease
* DSM-IV diagnoses or symptoms of substance use disorders, active within the last 60 days
* A score of 3 or higher on the suspiciousness/paranoia item of the Brief Psychiatric Rating Scale (BPRS)
* Acute, clinically significant gastrointestinal symptoms, such as nausea, vomiting, abdominal pain, diarrhea, melena, or hematochezia
* History of significant gastrointestinal disease or major gastrointestinal surgery
* Clinical instability of any kind that, in the investigator's opinion, could preclude safe participation in the study
* Known allergies that could preclude safe participation in the study
* Current presence of an electronically active implanted medical device
* Participation in another medical device study, or on any investigational drug or device within the last 30 days
* Inability to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Kane, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Zucker Hillside Hospital, Glen Oaks, New York

REFERENCES:
- [Result] Kane JM, Perlis RH, DiCarlo LA, Au-Yeung K, Duong J, Petrides G. First experience with a wireless system incorporating physiologic assessments and direct confirmation of digital tablet ingestions in ambulatory patients with schizophrenia or bipolar disorder. J Clin Psychiatry. 2013 Jun;74(6):e533-40. doi: 10.4088/JCP.12m08222. PMID 23842023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digital Health Feedback System (DHFS)
Started | 28
Completed | 27
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Digital Health Feedback System (DHFS)
Number analyzed (Participants) | 28
Age, Customized [Mean (Standard Deviation); unit: years] | 42.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Type of Mental Health Disorder [Count of Participants; unit: Participants]
  Bipolar Disorder | 12
  Schizophrenia | 16

OUTCOME MEASURES:

1. Primary Outcome: Positive Detection Accuracy
Description: Comparison of the detection rate of sensor-enabled placebo tablet ingestion using wireless observation (wirelessly observed therapy) to directly observed ingestion. Positive detection accuracy (PDA) for wirelessly observed therapy defined as the number of sensor ingestions detected by wireless observation, divided by the number confirmed ingestions using direct observation. PDA summarized as mean and 95% confidence interval.
Time Frame: 4 weeks
Population: 28 individuals with bipolar disorder (12) or schizophrenia (16)
Measure: Mean (95% Confidence Interval); unit: percentage of observed ingestions
Groups:
- Digital Health Feedback System (DHFS): Ingestion Sensor,...
Arm/Group | Digital Health Feedback System (DHFS)
Number analyzed (Participants) | 28
percentage of observed ingestions | 94 [85.4 to 100]

2. Secondary Outcome: System Safety
Description: Characterize, using summary (descriptive) statistics, the incidence and nature of system-related adverse events (AEs) and serious adverse events (SAEs) that are reported by study investigators over the course of the study
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Taking and Scheduling Adherence
Description: Characterize, using summary (descriptive) statistics, medication-taking behavior in free-living environment. Taking adherence defined as the number of ingestion sensors detected by the DHFS in the free-living environment, divided by the prescribed (planned) number of ingestions. Scheduling adherence defined as number of ingestion sensors detected by the DHFS within a ± 2-hour time window around the prescribed (planned) dosing time, divided by the total number of ingestion sensors detected by the DHFS.
Time Frame: 4 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Biometrics
Description: Characterize, using summary (descriptive) statistics, heart rate and rest/activity patterns in a free-living environment. Activity defined as the number of hours per day with recorded a recorded step rate ≥ 60 steps per minute
Time Frame: 4 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Usability
Description: Characterize, using summary (descriptive) statistics, the use of the digital health feedback system and its components by patients, caregivers, and healthcare providers. Use captured utilizing numeric scores collected from a standardized instrument, focusing on overall comfort and ease of DHFS use.
Time Frame: 4 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: User Experience
Description: Feedback and suggestions from patients, caregivers, and healthcare providers regarding system metrics and summary presentations of medication-taking, biometrics, and activities of daily living. Feedback includes free text and descriptive statistics summarizing numeric scores collected from a standardized instrument focusing on overall satisfaction with the DHFS and its components.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Digital Health Feedback System (DHFS): DHFS
Arm/Group | Digital Health Feedback System (DHFS)
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 6/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Health Feedback System (DHFS) (N=28)
schizoaffective disorder (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Health Feedback System (DHFS) (N=28)
Self-limited rash (Skin and subcutaneous tissue disorders) | 6 (9) — Nine non-serious AEs were reported by 6 subjects. All of the device-related, non serious AEs were characterized as skin irritation at the adhesive monitor placement location. The skin-related adverse events were mild in nature and self-limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No